CLINICAL TRIAL: NCT02924896
Title: The Chemical Structure of a Lipid Determines Its Effect on Blood Lipid Profile and Appetite Regulation
Brief Title: Effect of Palm Olein Intake on Lipid Profile and Appetite Regulation
Acronym: APO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16/WA/0117
Record Dates: First submitted 2016-09-28; First posted 2016-10-05 (Estimated); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Lipidaemia
Keywords: palm oil; apetite regulation
MeSH Terms: conditions — Hyperlipidemias | interventions — Soybean Oil

STUDY DESIGN:
Intervention Model Description: Number of participants 12
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Other): Palm Olein
  Interventions: Dietary Supplement: Palm olein; Dietary Supplement: Interesterified palm olein; Dietary Supplement: Soybean oil
- Arm 2 (Other): Soybean Oil
  Interventions: Dietary Supplement: Palm olein; Dietary Supplement: Interesterified palm olein; Dietary Supplement: Soybean oil
- Arm 3 (Other): Interesterified Palm Olein
  Interventions: Dietary Supplement: Palm olein; Dietary Supplement: Interesterified palm olein; Dietary Supplement: Soybean oil

INTERVENTIONS:
Dietary Supplement: Palm olein — 60g of palm olein will be given in a milkshake at breakfast
Dietary Supplement: Interesterified palm olein — 60g of interesterified palm olein will be given in a milkshake at breakfast
Dietary Supplement: Soybean oil — 60g of soybean oil will be given in a milkshake at breakfast

SUMMARY:
Aims: To investigate whether acute ingestions of palm oil will have an effect on appetite regulation

DETAILED DESCRIPTION:
Design: A randomized, single blind, cross over design including 4 single study visits separated by a week. Visit 1 is an acclimatization visit followed by visit 2,3, and 4 where different types of fat will be given.

Population: 12 healthy males and females aged between 18 and 60 years with body mass index (BMI) between 18.5- 29.9kg/m2 and normal fasting plasma glucose and no evidence of insulin resistance will be recruited. No-pre existing morbidity including cardiac, hepatic or renal disease, history of diabetes, hypertension or hyperlipidaemia.

Treatment: Acclimatization visit: At visit 1, all participants will be given a milkshake like drink containing fat, protein and carbohydrate. A cannula will be inserted for the duration of the study day but no blood will be taken. Studies show than during the first visit stress response can affect the metabolic response to the study drink resulting in inaccurate results.

Study visit 2,3,4: following the acclimatization visit, participants will attend 3 more study visits separated by a week to test the metabolic response to the following fats: palm olein, interesterified palm olein and soybean oil in random order. Participants will be asked to complete a visual analogue scale questionnaire about their appetite at each time point. Fasting and postprandial plasma glucose, insulin, appetite hormones and lipids will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and overweight male and female volunteers of all ethnicities (body mass index (BMI) of 18.5-29.9 kg/m2)
* Age between 18-60 years (inclusive)

Exclusion Criteria:

* Abnormal liver function test (elevated alanine aminotransferase and aspartate transaminase)/ abnormal kidney function test (elevated plasma creatinine)
* History of type 2 diabetes mellitus, cancer, stomach ulcers, drug abuse or alcoholism, gastrointestinal disorders like Crohn's disease
* Smokers
* On lipid/blood pressure- lowering medication/supplements
* Blood pressure>140/90 mm Hg
* Fasting total cholesterol > 6.2 mmol/L
* Fasting triacylglyceride > 2.0 mmol/L
* Subject must not be allergic to intervention
* Pregnancy and breastfeeding (pregnancy test will be undertaken at the screening visit)
* Subjects taking nutritional supplements or on any weight-loss programs
* Subjects who gained or lost ≥ 3kg weight in the past three months
* Subjects with history of hypo- and hyperthyroidism
* Subjects who are anaemic and those who donated blood within three months of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Research Facility official web page — http://imperial.crf.nihr.ac.uk/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Crossover study design where 12 participants will consume each of the three study oils at different sequence
Groups:
- Group Randomisation: Palm Olein, Soybean Oil, Interesterified Palm Olein
Period: First Intervention Day 1
Arm/Group | Group Randomisation
Started | 12
Completed | 12
Not Completed | 0
Period: Wash Out 7 Days
Arm/Group | Group Randomisation
Started | 12
Completed | 12
Not Completed | 0
Period: Second Intervention Day 1
Arm/Group | Group Randomisation
Started | 12
Completed | 12
Not Completed | 0
Period: Wash Out 7 Days
Arm/Group | Group Randomisation
Started | 12
Completed | 12
Not Completed | 0
Period: Third Intervention
Arm/Group | Group Randomisation
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Volunteers: Variables Male Female Combined n 12 Age (years) 35.7 (SD 18-60) Body Weight (kg) 66.6 (SD 11.5) BMI (kg/m2) 23.1 (SD 2.2)
  % Body Fat 24.5 (SD 8.9) Systolic Blood Pressure (mmHg) 114 (SD 10.5) Diastolic Blood Pressure (mmHg) 63 (SD 6.8) Heart Rate 74 (SD8.1)
Arm/Group | All Volunteers
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12
Age [Mean (Full Range); unit: years] | 35.7 [18 to 60]
Body Weight [Mean (Standard Deviation); unit: kilograms] | 66.6 (11.5)
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.1 (2.2)
% Body Fat [Mean (Standard Deviation); unit: percentage] | 24.5 (8.9)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 114 (10.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 63 (6.8)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 74 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Appetite Hormones PYY
Description: blood samples will be collected at specific time points presented as minutes from consumption of mixed meal.
  time (minutes)=-15, -5, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420, 480.
Time Frame: 480 minutes
Population: The AUC it is estimated across the timepoints above and across the different number of patients per arm.
Measure: Mean (Standard Deviation); unit: mmol/L*min
Groups:
- Soybean: Soybean oil: 60g of soybean oil will be given in a milkshake at breakfast
- Palm Oil: Palm olein: 60g of palm olein will be given in a milkshake at breakfast
Arm/Group | Soybean | Palm Oil | Interesterified Palm Olein
Number analyzed (Participants) | 12 | 12 | 12
mmol/L*min | 58.5 (11.3) | 60 (12.1) | 56 (10.5)

2. Secondary Outcome: Change From Baseline in Glucose,
Description: as for outcome 1
Time Frame: 480 min
Population: The AUC it is estimated across the timepoints above and across the different number of patients per arm.
Measure: Mean (Standard Deviation); unit: mmol/L*min
Groups:
- Soya: Soya milk shake
- Palm Oil: Palm oil milk shake
- Palm Ol: Interesterified Palm Olein
Arm/Group | Soya | Palm Oil | Palm Ol
Number analyzed (Participants) | 12 | 12 | 12
mmol/L*min | 1400 (250) | 1545 (240) | 1486 (230)

3. Secondary Outcome: Change From Baseline in Appetite Hormones GLP_1
Description: Change From Baseline in Appetite Hormones
  Hide Description:
  blood samples will be collected at specific time points presented as minutes from consumption of mixed meal.
  time (minutes)=-15, -5, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420, 480.
Time Frame: ime (minutes)=-15, -5, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420, 480. Time Frame: 480 minutes
Measure: Mean (Standard Error); unit: mmol/L*min
Arm/Group | Soybean | Palm Oil | Interesterified Palm Olein
Number analyzed (Participants) | 12 | 12 | 12
mmol/L*min | 43.8 (12.7) | 32 (10) | 55 (14.1)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: No difference
Groups:
- Palm Olein: palm olein: 60g of interesterified palm olein will be given in a milkshake at breakfast
- Soya Bean: Soybean oil: 60g of soybean oil will be given in a milkshake at breakfast
Arm/Group | Palm Olein | Interesterified Palm Olein | Soya Bean
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT02924896/Prot_SAP_ICF_000.pdf